CLINICAL TRIAL: NCT03410836
Title: Impact of Intraoperative Intravenous Lidocaine Administered During Laparoscopic Colorectal Surgery on Remifentanil Consumption, Postoperative Pain and Immune Cell Activity: A Pilot Study
Brief Title: Impact of Intravenous Lidocaine During Colorectal Surgery on Pain and Immune Functions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Foundation of Anesthesia and Resuscitation of Quebec (Unknown)
Responsible Party: Principal Investigator, Philippe Richebe, Director of Research in Anesthesiology, MD, PhD, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-1066
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Intravenous Lidocaine and Immunity
Keywords: lidocaine; colorectal cancer; laparoscopy surgery; anesthesia; inflammation; cytokine; post-operative immunosuppression
MeSH Terms: conditions — Colorectal Neoplasms; Inflammation

STUDY DESIGN:
Intervention Model Description: Two groups of patients. Randomization into the treatment group or placebo group according to a randomization list for a total number of patients of 60.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drug administered intraoperatively (intravenous lidocaine or intravenous placebo) will be blinded to patient, anesthesiologist, research nurse for the entire duration of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous lidocaine (IVL) (Experimental): Will receive during the colorectal surgery under General Anesthesia intravenous lidocaine bolus 1.5mg/kg at the beginning of anesthesia (induction) and 1.5mg/kg/h until the end of anesthesia.
  Interventions: Drug: intravenous lidocaine (IVL)
- Placebo (Placebo Comparator): Will receive the same volume of normal saline for the entire duration of anesthesia.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: intravenous lidocaine (IVL) — lidocaine 2% will be used for induction (1 syringe of 5 ml, administered dose of 1.5 mg / kg) and for intra-operative infusion (1 syringe of 30 ml, infusion dose of 1.5 mg / kg / h). Lidocaine syringes and placebo will be prepared on a blinded manner so that the investigating anesthesiologist in charge of the patient in the operating room, as well as the respiratory therapist and the recovery room nurse and the floors do not know what the patient received during the anesthesia (whether IVL or placebo).
  Arms: intravenous lidocaine (IVL)
Other: Placebo — Group Control will receive (double blinded) an infusion of saline at the same volume and regimen than the lidocaine 2% group (IVL).
  Arms: Placebo

SUMMARY:
This study evaluates the impact of intraoperative intravenous lidocaine administered during laparoscopic colorectal surgery on the intraoperative remifentanil consumption as well as postoperative pain and opioid requirements. It will evaluate immune cell activity for 48hours after surgical stress and general anesthesia with or without intravenous lidocaine.

DETAILED DESCRIPTION:
Hypothesis: We hypothesize that the intravenous lidocaine (IVL) versus placebo administered during laparoscopic colorectal surgery will allow for: a reduction in intraoperative remifentanil consumption, an improvement in patients' early rehabilitation after surgery, and an enhancement of the immune profile of our patients through an increase in the balance Th1/Th2 and cellular immunity.

Background: so far, IVL was shown to have several properties: analgesic, anti-inflammatory, and anti-hyperalgesic. Its effects on rehabilitation and pain are still controversial except for abdominal surgery. To date, no study evaluated the impact of IVL in colorectal surgery on intraoperative consumption of remifentanil. Postoperative immune suppression is multifactorial and depends on the surgical traumatism, but also on the doses of opioids given during anesthesia. No study evaluated in colorectal surgery the impact of IVL on postoperative cellular immunity and on the risk of cancer recurrence.

Specific Objectives: primary objective: to reduce by 30% the consumption of remifentanil in the IVL group versus the placebo group; secondary objectives: to evaluate the quality of recovery from anesthesia in the OR (awakening and extubation time), in the PACU and on the wards (pain scores, opioid consumption with patient controlled analgesia (PCA), postoperative nausea and vomiting (PONV), transit recovery time, time in PACU and time in hospital), and to evaluate the postoperative inflammatory parameters and adaptative immune functions (Th1/Th2) until postoperative 48h.

Methods: 60 adult patients ASA 1-3 scheduled for elective laparoscopic colorectal surgery will be included in this randomized controlled trial. Randomisation will be into group Control (C) and Lidocaine (IVL). Anesthesia and monitoring will be standardized and accompanied with the monitoring of the depth of anesthesia (BISpectral index, Medtronic) and the depth of analgesia (NoL index, Medasense LTD, recorded on an observational manner). IVL group will blindly be administered intravenous 1.5 mg/kg lidocaine bolus and then 1.5 mg/kg/h until the end of the surgery as previously described. C group will receive the same amount (ml) of placebo. Statistics: a preliminary analysis (idem group C) showed that the total amount of remifentanil given for this type of surgery was 2481+/-985 mcg (duration 141+/-30Min). Considering that we wish to reduce by 30% the remifentanil consumption in the group IVL, the number of patients to be included per group is 30 (alpha 0.05 and beta 20%).

Significance/Importance: this study will evaluate the impact of IVL on intraoperative consumption of remifentanil but also on immune functions after surgery in order to reduce the risk of cancer recurrence. If this study brings positive results, this will lead to a significant change in clinical practice of anesthesia. This is a pilot study on the immune functions, but this might bring very strong results to ask for future grants on the impact of IVL on cancer recurrence.

Study Design: Prospective, randomized controlled study. Subject Population: Adult patients scheduled to undergo elective laparoscopic colorectal surgery under general anesthesia.

Sample Size: 60 patients will be evaluated in this study. Study Duration: 1 year. Study Center: Maisonneuve-Rosemont Hospital, CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada.

Adverse Events: None expected.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I, II or III
* Patients older than 18 years
* Colonic surgery
* Classical management of ERAS program patients in our center

Exclusion Criteria:

* Arrhythmia, abnormal electrocardiographic , antiarrhythmic therapy
* Immunosuppressive treatments, corticosteroids or long-term NSAIDs (multiple weekly doses) or during preoperative 48 hours
* conversion intraoperative of a laparoscopic surgical technique to a laparotomy technique
* Pregnant women
* Inability to complete the questions related to this study
* Inability to use hydromorphone postoperative PCA
* Intolerance or allergy to lidocaine, hydromorphone or any other drug that is included in the protocol for perioperative management

Unexpected events leading to the exclusion:

* Difficult unplanned intubation
* Surgical complication requiring aggressive haemodynamic support (vasopressors, inotropes, transfusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of total intraoperative remifentanil consumption by 30% in the intravenous lidocaine ("IVL") group compared with the control group ("C"). Total consumption of remifentanil in mcg. | Intra-operative, 5 hours
  Reduction of total intraoperative remifentanil consumption by 30% in the intravenous lidocaine group compared with the control group.

SECONDARY OUTCOMES:
Evaluation of the number of remifentanil boluses given intraoperatively (n) | T0 to end of surgery, 5 hours
  Evaluation of the number of remifentanil boluses given intraoperatively, based on the intraoperative NOL index from T0 which is the time of the incision
Assessment of total consumption of inhaled anesthetic desflurane in ml | intra-operative
  The Dräger Perseus A500 that we have in each anesthesia room offers the opportunity to get the ml of halogenous gas consumed precisely, and our electronic extraction database will allow to have this data in ml per second and the total at the end of surgery
Evaluation of time for extubation | post-operative 1 hour
  Evaluation of time for extubation after surgery in the operating room
Evaluation of the hydromorphone dose in mg used in the post-operative care unit (PACU) titration | in recovery room, 3 hours
  Evaluation of the hydromorphone dose in mg used as post-operative titration immediately in the recovery room (PACU) to obtain NRS pain scores < 3/10
Evaluation of the nausea and vomiting scores, 0 to 3 scale | 48 hours
  Evaluation of the nausea and vomiting scores (0 to 3) for the first 48 hours
Evaluation of the length of stay in the recovery room based on the Aldrete scores (Score from 0 to 9) | in recovery room, 3 hours
  Evaluation of the length of stay in the recovery room based on the Aldrete scores (time to be ready to leave the recovery room)
total hydromorphone consumption (mg) after PACU, on wards | 48 hours
  total hydromorphone consumption (mg given by Patient Controlled Analgesia) on wards for 48 hours
Evaluation of the satisfaction of the patient scale 0 to 100 (%) | 48 hours postoperatively
  Evaluation of the satisfaction of the patient as for the management of his pain for 48 hours
Assessment of total hospital duration of stay in hours | 7 days postoperatively
  Assessment of total hospital stay in hours
Evaluation of the time in hours required for the emission of a first gas in hours | 5 days postoperatively
  Evaluation of the time in hours required for the emission of a first gas, a sign of resumption of normal intestinal function
Assessment of rehabilitation scores and cognitive functions | 2 days
  Assessment of rehabilitation scores and cognitive functions at 48h after surgery
Assessment of cytokines in plasma | 48 hours
  Assessment of inflammation parameters by blood sample for 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Richebé, MD, PhD, Principal Investigator — CIUSSS Est de l'ile de Montreal
Locations (1):
- Hôpital Maisonneuve-Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No